CLINICAL TRIAL: NCT04618614
Title: The Effect of High-definition Transcranial Direct Current Stimulation of the Somatosensory Area on Upper Limb Motor Performance in Healthy Adults
Brief Title: The Effect of Transcranial Direct Current Stimulation of the Somatosensory Area on Upper Limb Motor Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ariel University (Other)
Collaborators: Tel Aviv University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AU-HEA-SFT-20190326-B
Record Dates: First submitted 2020-11-01; First posted 2020-11-06 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2021-01

CONDITIONS: Healthy
Keywords: transcranial direct current stimulation, motor performance

STUDY DESIGN:
Intervention Model Description: randomized controlled trial (RCT)
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HD-tDCS S1 1 mA (Experimental): Single session of 15-min HD-tDCS to the right primary somatosensory cortex with an intensity of 1 mA. The session will last approximately one hour.
  Interventions: Device: HD-tDCS 1 mA to S1
- HD-tDCS M1 1 mA (Active Comparator): Single session of 15-min HD-tDCS to the right primary motor cortex with an intensity of 1 mA. The session will last approximately one hour.
  Interventions: Device: HD-tDCS 1 mA to M1
- Sham control (Sham Comparator): Single session of 15-min HD-tDCS to the right primary somatosensory cortex with an intensity of 1 mA. The session will last approximately one hour.
  Interventions: Device: Sham control

INTERVENTIONS:
Device: HD-tDCS 1 mA to S1 — Anodal high definition transcranial direct current stimulation of the right primary somatosensory cortex with an intensity of 1 mA
  Arms: HD-tDCS S1 1 mA
Device: HD-tDCS 1 mA to M1 — Anodal high definition transcranial direct current stimulation of the right primary motor cortex with an intensity of 1 mA
  Arms: HD-tDCS M1 1 mA
Device: Sham control — Sham stimulation of the right primary somatosensory cortex
  Arms: Sham control

SUMMARY:
to investigate the effect of transcranial direct current stimulation of the somatosensory area on upper limb motor performance in healthy adults

DETAILED DESCRIPTION:
60 healthy subjects will be randomly allocated to one of three groups: (a) 15- min of High-Definition transcranial direct current stimulation (HD-tDCS) on primary somatosensory cortex (S1) with an intensity of 1 milliampere (mA) (HD-tDCS S1); (b) 15-min of HD-tDCS on primary motor cortex (M1) with an intensity of 1 mA (HD-tDCS M1); and (c) 15-min of sham HD-tDCS (HD-tDCS sham).

The stimulation will be administered noninvasively using an M x N 9-channel high definition transcranial electrical current stimulator from Soterix Medical (New York, NY). In the HD-tDCS S1 group, the anodal stimulation will target the right postcentral gyrus. In the HD-tDCS M1 group, the anodal stimulation will target the right primary motor cortex (brodmann area 4). The location of the electrodes will be placed based on HD-Targets brain modelling software (Soterix Medical, New York, NY).

Tests (motor and sensory tasks): The non-dominant left arm will be tested. Motor task: The subjects will perform a sequential point-to-point movement task on the graphics tablet. Initially, the participants will be required to perform 3 sequences without errors to familiarize themselves with the setup, the task and the sequence. Then, they will perform the pre-test which consists of two blocks of 6 sequences, i.e. 12 sequences, with a 30 s break between blocks. Two min after starting the appropriate stimulation, they will perform 2 blocks of 6 sequences (identical to the pre-test). After finishing the tDCS stimulation, the participants will perform a post-test, which is also identical to the pre-test. Three outcome measures will be used: movement time (s), reaction time (s) and straight line deviation (cm) of the reaching movements. Sensory tasks: discriminative task (two point orientation discrimination) and proprioception task will be included. The sensory tasks will be performed with eyes blindfolded. In the discriminative task the experimenter will deliver a stimuli by a two-pronged instrument at intervals of 2,3,4,5 mm to the distal phalanx of fingers 2 and 5 of the left hand. The stimulus will be oriented either across or down (total of 16 stimuli). Subjects will be asked to Identify the orientation of the stimulation. The outcome measure will be the percentage of correct answers. In the proprioceptive task, the subjects will perform a one direction point-to-point (target) movement task on the graphics tablet. The task will include 20 movements, 10 passive movements and 10 active movements. After every passive movement with eyes blindfolded, the subject will be asked to perform a similar active movement. Initially, the participants will be asked to perform four movements to familiarize themselves with the setup (the first two movements will be passive and active movements with eyes open, and the following two movements will be passive and active movements with eyes blindfolded). The outcome measure will be the end point error (cm) which is the distance between the target and the actual arrival location.

ELIGIBILITY:
Inclusion Criteria:

* aged between 20 and 35
* right-hand dominant
* healthy according to self report

Exclusion Criteria:

* taking psychiatric medications
* a history of drug / alcohol abuse or dependence
* psychiatric or neurological disorder
* a history of seizures
* metal implants in their head
* musculoskeletal deficits interfering with task performance (proper reaching performance in sitting)

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-11-10 (Actual); Primary Completion 2021-01-07 (Actual); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in movement time (s) from baseline to intervention | Baseline (immediately before stimulation), two minutes after starting the stimulation
  Time from movement onset (first time the tangential velocity was greater than 5% of the peak tangential velocity) until the end of the movement (the last time the tangential velocity will be greater than 5% of the peak tangential velocity). Improved motor performance will be indicated by a shorter movement time.
Change in movement time (s) from baseline to posttest | Baseline (immediately before stimulation), immediately post stimulation
  Time from movement onset (first time the tangential velocity was greater than 5% of the peak tangential velocity) until the end of the movement (the last time the tangential velocity will be greater than 5% of the peak tangential velocity). Improved motor performance will be indicated by a shorter movement time.
Change in movement time (s) from intervention to posttest | Two minutes after starting the stimulation, immediately post stimulation
  Time from movement onset (first time the tangential velocity was greater than 5% of the peak tangential velocity) until the end of the movement (the last time the tangential velocity will be greater than 5% of the peak tangential velocity). Improved motor performance will be indicated by a shorter movement time.
Change in reaction time (s) from baseline to intervention | Baseline (immediately before stimulation), two minutes after starting the stimulation
  Time between when the target appeared in green (changed color from white to green), and movement onset. Improved motor performance will be indicated by a shorter reaction time.
Change in reaction time (s) from baseline to posttest | Baseline (immediately before stimulation), immediately post stimulation
  Time between when the target appeared in green (changed color from white to green), and movement onset. Improved motor performance will be indicated by a shorter reaction time.
Change in reaction time (s) from intervention to posttest | Two minutes after starting the stimulation, immediately post stimulation
  Time between when the target appeared in green (changed color from white to green), and movement onset. Improved motor performance will be indicated by a shorter reaction time.
Change in straight line deviation (cm) from baseline to intervention | Baseline (immediately before stimulation), two minutes after starting the stimulation
  Path deviation from a straight line (zero means no deviation). Improved motor performance will be indicated by a shorter deviation.
Change in straight line deviation (cm) from baseline to posttest | Baseline (immediately before stimulation), immediately post stimulation
  Path deviation from a straight line (zero means no deviation). Improved motor performance will be indicated by a shorter deviation.
Change in straight line deviation (cm) from intervention to posttest | Two minutes after starting the stimulation, immediately post stimulation
  Path deviation from a straight line (zero means no deviation). Improved motor performance will be indicated by a shorter deviation.

SECONDARY OUTCOMES:
Change in the correct answers (%) of discriminative task from baseline to posttest | Baseline (immediately before stimulation), immediately after the motor posttest
  Identification of the orientation of the stimulus. Improved sensation will be indicated by a higher % of correct answers.
Change in end point error (cm) of proprioception task from baseline to posttest | Baseline (immediately before stimulation), immediately after the motor posttest
  The distance between the target point to the actual arrival location. Improved sensation will be indicated by a smaller distance.

CONTACTS AND LOCATIONS:
Overall Officials: Silvi Frenkel-Toledo, PhD, Principal Investigator — Ariel University
Locations (1):
- Ariel University, Ariel, Israel

IPD SHARING:
Plan to Share IPD: No
The datasets (Study Protocol, Statistical Analysis Plan, Informed Consent Form, Analytic Code generated during and/or analyzed during the current study) will be available from the corresponding author on reasonable request.